CLINICAL TRIAL: NCT00230035
Title: A Randomized, Open Label, Phase II Multicenter Study of Non-Myeloablative Autologous Transplantation With Auto-CD34+HPC Versus Currently Available Immunosuppressive/Immunomodulatory Therapy for Treatment of Systemic Lupus Erythematosus
Brief Title: Lupus Immunosuppressive/Immunomodulatory Therapy or Stem Cell Transplant (LIST)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Recommended by DSMB due to lack of accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT SCSLE-01
Record Dates: First submitted 2005-09-28; First posted 2005-09-30 (Estimated); Last update posted 2013-02-01 (Estimated); Status verified 2013-01

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Leukapheresis; Plasmapheresis; Antilymphocyte Serum; Methylprednisolone; Granulocyte Colony-Stimulating Factor; Adrenal Cortex Hormones; Mycophenolic Acid; Azathioprine; Immunoglobulins, Intravenous; Methotrexate; Rituximab; Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): high dose immunosuppressie therapy (HDIT) followed by HSCT (hemopoietic stem cell transplantation).
  Interventions: Procedure: Leukapheresis; Procedure: Non-myeloablative high dose immunosuppressive therapy conditioning (HDIT); Procedure: Autologous CD34+HPC transplantation (HSCT)
- 2 (Active Comparator): Currently available immunosuppressive/immunomodulatory therapy
  Interventions: Procedure: Plasmapheresis; Drug: Rabbit anti-thymocyte globulin; Drug: Methylprednisolone; Drug: Growth colony stimulating factor (G-CSF); Drug: Corticosteroids; Drug: Mycophenolate mofetil; Drug: Azathioprine; Drug: Intravenous immunoglobulin; Drug: Methotrexate; Drug: Rituximab; Drug: Leflunomide

INTERVENTIONS:
Procedure: Leukapheresis
  Arms: 1
Procedure: Non-myeloablative high dose immunosuppressive therapy conditioning (HDIT)
  Arms: 1
Procedure: Autologous CD34+HPC transplantation (HSCT)
  Arms: 1
Procedure: Plasmapheresis
  Arms: 2
Drug: Rabbit anti-thymocyte globulin
  Arms: 2
Drug: Methylprednisolone
  Arms: 2
Drug: Growth colony stimulating factor (G-CSF)
  Arms: 2
Drug: Corticosteroids
  Arms: 2
Drug: Mycophenolate mofetil
  Arms: 2
Drug: Azathioprine
  Arms: 2
Drug: Intravenous immunoglobulin
  Arms: 2
Drug: Methotrexate
  Arms: 2
Drug: Rituximab
  Arms: 2
Drug: Leflunomide
  Arms: 2

SUMMARY:
Systemic lupus erythematosus, also known as lupus or SLE, is a chronic, multisystem, autoimmune disease in which the body's internal system of defense attacks its own normal tissues. This abnormal autoimmune response can result in damage to many parts of the body, especially the skin, joints, lungs, heart, brain, intestines, and kidneys. Both genetic and environmental risk factors are involved in the development of lupus, but these are poorly understood.

SLE has an overall 10-year survival between 80 and 90%. However, we estimate that severe lupus not responding to the usual available treatments has a 50% mortality rate in 10 years. Kidney problems occur in 30% to 50% of lupus patients and may progress to kidney failure. Kidney disease due to lupus occurs more frequently in African-Americans and Hispanics. Lupus can affect many parts of the body and cause damage, but the severe form can result in death from kidney disease; cardiovascular disease, specifically atherosclerosis; central nervous system disease; and infections.

Currently, no single standard therapy for treatment of severe SLE exists. Usually physicians prescribe an aggressive regimen of one or a combination of immunosuppressive/immunomodulatory treatments. This approach to therapy for all forms of severe SLE derives largely from studies of lupus nephritis. Current treatment, although effective in many people, are not effective in all patients and are associated with drug-induced morbidity. The design of the control arm for this study reflects the current status of treatment of SLE in the academic setting. Investigators may choose from a list of commonly used and currently available immunosuppressive/immunomodulatory treatments to optimize the treatment of their patients, based on their past treatment history and response to those treatments. Study treatments may consist of corticosteroids, cyclophosphamide (CTX), azathioprine, methotrexate, cyclosporine, mycophenolate mofetil (MMF), plasmapheresis, intravenous immunoglobulin (IVIG), rituximab, and leflunomide. Treatment may be changed as frequently and as necessary within the first year of the study to control the manifestations of SLE in each patient. New therapies that become available during the course of this trial may be added to the list of approved medications for this study.

In response to the absence of a uniformly effective treatment for severe lupus, autologous hematopoietic stem cell transplantation (HSCT) has been proposed as a potential therapy. Hematopoietic stem cells are immature blood cells that can develop into all of the different blood and immune cells the body uses. Researchers believe that resetting the immune system may stop or slow down the progression of the disease. The main purpose of this study is to compare two ways of treating SLE: 1) high-dose immunosuppressive therapy (HDIT) followed by HSCT and 2) currently available immunosuppressive/immunomodulatory therapies.

DETAILED DESCRIPTION:
SLE is a chronic, multisystem, inflammatory autoimmune disease in which the body's immune cells wrongly attack its own tissues. It is defined by the presence of circulating antinuclear antibodies that are directed against nucleosomal DNA-histone complexes, native double-stranded DNA (dsDNA), small nuclear ribonucleoproteins (Sm and RNP), single-stranded DNA, and phospholipids moieties on platelets and other tissues, indicating a failure of the regulatory systems involved in maintenance of immunologic tolerance to self-antigens. Despite use of currently available therapies, patients experience relapses of their lupus. Over time, patients develop significant morbidity from the disease as well as from medications, including glucocorticoids, used for treatment. The main purpose of this study is to compare two ways of treating SLE: 1) high-dose immunosuppressive therapy (HDIT) followed by HSCT and 2) currently available immunosuppressive/immunomodulatory therapies.

1. One group of study participants will undergo autologous hematopoietic stem cell transplantation. With this treatment, they will first undergo mobilization, a process that removes hematopoietic stem cells from their blood. Then they will receive high doses of chemotherapy to suppress their abnormal immune systems, followed by the reintroduction of the purified stem cells to re-establish their immune systems.

   Medications are used to mobilize (i.e., encourage) blood cell precursors to multiply and move from the bone marrow to the bloodstream. These precursors (or autologous stem cells) can be harvested (collected) from the bloodstream during a process called apheresis and then transplanted (infused) back into the patient's body after chemotherapy has been given. HDIT can suppress the immune system, reducing the effectiveness or perhaps eliminating most of the immune cells that cause the progression of SLE. Autologous hematopoietic stem cell transplantation (HSCT) following HDIT hastens the return of the body's ability to produce blood cells. HDIT with HSCT has been identified as a potential treatment alternative to standard chemotherapy treatments.

   One group of study participants will undergo autologous hematopoietic stem cell transplantation. With this treatment, they will first undergo mobilization, a process that removes hematopoietic stem cells from their blood. Then they will receive high doses of chemotherapy to suppress their abnormal immune systems, followed by the reintroduction of the purified stem cells to re-establish their immune systems.

   Medications are used to mobilize (i.e., encourage) blood cell precursors to multiply and move from the bone marrow to the bloodstream. These precursors (or autologous stem cells) can be harvested (collected) from the bloodstream during a process called apheresis and then transplanted (infused) back into the patient's body after chemotherapy has been given. HDIT can suppress the immune system, reducing the effectiveness or perhaps eliminating most of the immune cells that cause the progression of SLE. Autologous hematopoietic stem cell transplantation (HSCT) following HDIT hastens the return of the body's ability to produce blood cells. HDIT with HSCT has been identified as a potential treatment alternative to standard chemotherapy treatments.

   Participants assigned to the first treatment group will undergo mobilization with CTX and granulocyte colony stimulating factor (G-CSF) beginning 2 weeks after randomization. In preparation for the transplant process. a central venous line (plastic tube) will be inserted into the neck or chest vein; this tube will be used to administer stem cells and medications and for drawing blood. IV CTX, followed by G-CSF, will be given injected under the skin beginning 3 days after CTX. G-CSF will be given for about 4 to 7 days, to boost the body's production of blood precursor cells. These precursor cells will be collected through the central venous line through apheresis. In this process, whole blood is collected through a needle in an arm vein and directed to a cell-separating machine, where the white cells are separated and saved. The rest of the blood is returned to the patient through the same needle. Several apheresis procedures will be required to collect enough cells for the autologous transplant.

   Within 3 weeks of the apheresis stem cell collection, the first group's participants will be admitted to the hospital and will undergo a five-day conditioning regimen consisting of IV CTX and rabbit anti-thymocyte globulin (rATG). This regimen will suppress the malfunctioning immune system and prepare the patient's body to receive the precursor cells previously collected during apheresis. The stem cells will be infused after the five-day conditioning regimen. The return of the precursor cells is called autologous stem cell transplantation. During the hospitalization a specialized team of transplant physicians and nurses will closely monitor the participants until their bone marrow recovers and the participants are well enough to be discharged. The hospital stay will be approximately 21 days after the autologous stem cell transplant. Upon discharge, the patient will return home and will follow-up at the treatment center at Weeks 1 and 3 post-transplantation for close monitoring by the transplant team. Participants will also be followed by the study rheumatologist monthly at the treatment center for 30 months.
2. The other group of study participants will receive immunosuppressive/immunomodulatory therapy as prescribed by the study rheumatologist, based on the organ systems affected and prior treatment history. Therapy may include one or a combination of the following treatments: corticosteroids, azathioprine, methotrexate, cyclosporine, MMF, plasmapheresis, IVIG, rituximab, and leflunomide. As new drugs become available and a part of the usual medications for the treatment of SLE, they may be approved for use in this study. Treatment may be changed as frequently as necessary within the first year of the study to control the manifestations of SLE in each patient. Treatment for the second group will begin 1 week after randomization; patients will be seen monthly at the treatment center for 30 months.

Corticosteroid dosage tapering will be monitored closely; the schedule for tapering will be the same in both groups. To reduce the possibility of disease flare. a slow tapering of 10% per month will occur for the first six months. Tapering will continue in a prescribed manner to achieve a dose equivalent of 10 mg/day of prednisone or less by one year post-treatment.

All participants will have monthly follow-up visits for 30 months after treatment has been initiated. Study visits will include a physical exam, clinical assessments, rheumatology evaluations, and blood and urine collections. Participants will be asked to complete questionnaires assessing their lupus disease. Neuropsychiatric assessments, echocardiogram, CT scan of brain, renal biopsy, pulmonary function test, dual-energy x-ray absorptiometry scan (DEXA scan), magnetic resonance imagery scan, electromyograph scan (EMG), bone marrow biopsy and aspiration and lumbar puncture may occur at selected visits, based on each individual's manifestations of lupus and clinical indication. Participants will also receive certain vaccinations at selected visits. Participants will be contacted by phone each and every week throughout the study. There will be an extension period for those patients that have completed their treatment and follow-up visits during the study's 5-year duration. Participants will be contacted via telephone, e-mail, or visit every 3 months to assess their use of concomitant medications and immunosuppressive/immunomodulatory therapy and corticosteroids.

Five treatment centers across the United States, all leaders in the fields of transplantation and rheumatology, are participating in this research study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between the ages of 18 and 60 years, inclusive
* Meet at least 4 of 11 American College of Rheumatology (ACR) Revised Classification Criteria for SLE
* Have at least one of the following conditions defining severe steroid refractory disease:

  a) Lupus nephritis - Subjects must have severe disease, defined as meeting criteria for BILAG renal category A, and be corticosteroid dependent while receiving at least 6 months of pulse CTX at doses of 500 to 1000 mg/m2 every 4 weeks or MMF at of 2 g/day or greater. If nephritis is to constitute the sole eligibility, a renal biopsy performed within 11 months of the date of screening must show ISN/RPS 2003 classification of lupus nephritis Class III or IV disease. A renal biopsy must demonstrate the potential of a reversible (non-fibrotic) component. b) Visceral organ involvement other than nephritis - Subjects must be without mesenteric vasculitis. The subject must be BILAG cardiovascular/respiratory category A, vasculitis category A, or neurologic category A, and be corticosteroid dependent while receiving at least 3 months of oral (2 to 3 mg/kg/day or greater) or IV CTX (500 mg/m2 or greater every 4 weeks). c) Cytopenias that are immune-mediated - Subjects must be BILAG hematologic category A and be corticosteroid dependent while receiving at least one of the following: azathioprine at 2 mg/kg/day or greater for at least 3 months, MMF at 2 g/day or greater for more than 3 months, CTX at 500 mg/m2 or greater intravenously every 4 weeks or 2 mg/kg/day orally for at least 3 months, cyclosporine at 3 mg/kg/day or greater for at least 3 months, or have had a splenectomy. d) Mucocutaneous disease - Subjects must meet BILAG mucocutaneous category A and be corticosteroid dependent while receiving at least 1 of the following: azathioprine at 2 mg/kg/day or greater for at least 3 months; methotrexate at 15 mg/week or greater for at least 3 months; CTX at 500 mg/m2 or greater intravenously every 4 weeks or 2 mg/kg/day or greater orally for at least 3 months, cyclosporine at 3 mg/kg/day or greater for at least 3 months, or MMF at doses 2 g/day or greater for at least 3 months. e) Arthritis/myositis - Subjects must meet BILAG musculoskeletal category A and be corticosteroid dependent while receiving at least one of the following: azathioprine at 2 mg/kg/day or greater for at least 3 months, methotrexate at 15 mg/week or greater for at least 3 months, CTX at 500 mg/m2 or greater intravenously every 4 weeks or 2 mg/kg/day or greater orally for at least 3 months, MMF at 2 g/day or greater for at least 3 months, or cyclosporine at 3 mg/kg/day or greater for at least 3 months.
* Have the ability and willingness to provide written informed consent. In case of lupus cerebritis, a person designated by the subject may give consent.
* Must be ANA positive

Exclusion Criteria:

* HIV positive status
* Any active systemic infection
* Hepatitis B surface antigen positive
* Hepatitis C PCR positive
* Use of immunosuppressive agents for other indications other than SLE
* Any comorbid illness that in the opinion of the investigator would jeopardize the ability of the subject to tolerate therapy
* For lupus nephritis: renal biopsy, performed within 11 months of the screening date, showing Class I, II, or V disease or Class III or IV disease in conjunction with total sclerosis of 50% or more of the glomeruli
* Ongoing cancer. Patients with localized basal cell or squamous skin cancer are not excluded.
* Pregnancy, unwillingness to use acceptable means of birth control, or unwilling to accept or comprehend irreversible sterility as a side effect of therapy
* Psychiatric illness or mental deficiency not due to active lupus cerebritis making compliance with treatment or informed consent impossible
* Hemoglobin adjusted diffusion capacity test (DLCO) less than 30% at screening
* Resting left ventricular ejection fraction (LVEF) 40% or less as evaluated by echocardiogram
* History of an allergic reaction or hypersensitivity to Escherichia coli recombinant proteins, CTX, or any part of the investigative or control therapy
* SGOT/SGPT greater than 2 x the upper limit of normal, unless due to active lupus
* ANC 1000 or greater if not due to active SLE
* Subdural hematoma or any active intracranial bleeding documented within 30 days of the screening visit
* Failure to be approved for participation in this study by the SCSLE Protocol Eligibility Review Committee
* Positive tuberculin skin test
* Presence of mesenteric vasculitis

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09

PRIMARY OUTCOMES:
Mortality resulting from treatment, underlying disease, or unrelated causes | At Month 30

CONTACTS AND LOCATIONS:
Overall Officials: Richard Burt, MD, Study Chair — Division of Immunotherapy, Northwestern University; Bevra Hahn, MD, Study Chair — Division of Rheumatology, Department of Medicine, University of California, Los Angeles; Kenneth Kalunian, MD, Study Chair — Division of Rheumatology, Allergy, and Immunology, University of California, Los Angeles; Ann Traynor, MD, Study Chair — Division of Hematology and Oncology, University of Massachusetts Medical School; Keith Sullivan, MD, Study Chair — Division of Cellular Therapy, Department of Medicine, Duke University; Betty Diamond, MD, Study Chair — Department of Medicine, Columbia University
Locations (5):
- United States (5):
  - UCSD, Thornton Hospital, La Jolla, California
  - UCLA, Rehabilitation Center, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Feinstein Institute for Medical Research NS-LIJ Health System, Manhassat, New York
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Burt RK, Marmont A, Arnold R, Heipe F, Firestein GS, Carrier E, Hahn B, Barr W, Oyama Y, Snowden J, Kalunian K, Traynor A. Development of a phase III trial of hematopoietic stem cell transplantation for systemic lupus erythematosus. Bone Marrow Transplant. 2003 Aug;32 Suppl 1:S49-51. doi: 10.1038/sj.bmt.1703943. PMID 12931242
- [Background] Openshaw H, Nash RA, McSweeney PA. High-dose immunosuppression and hematopoietic stem cell transplantation in autoimmune disease: clinical review. Biol Blood Marrow Transplant. 2002;8(5):233-48. doi: 10.1053/bbmt.2002.v8.pm12064360.
- [Background] Traynor AE, Barr WG, Rosa RM, Rodriguez J, Oyama Y, Baker S, Brush M, Burt RK. Hematopoietic stem cell transplantation for severe and refractory lupus. Analysis after five years and fifteen patients. Arthritis Rheum. 2002 Nov;46(11):2917-23. doi: 10.1002/art.10594. PMID 12428232